CLINICAL TRIAL: NCT03283137
Title: A Phase I, Open-label, Dose-escalation Study to Assess the Safety, Tolerability and Efficacy of the Combination of Pembrolizumab With TGR-1202 in Patients With Relapsed/Refractory CLL and B-Cell Non-Hodgkin Lymphoma (NHL)
Brief Title: Combination of Pembrolizumab With TGR-1202 in Patients With Relapsed/Refractory CLL and B-cell NHL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-0901
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: CLL; B-cell Non Hodgkin Lymphoma
Keywords: CLL; B-cell Non Hodgkin Lymphoma; pembrolizumab; TGR-1202
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — umbralisib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- TGR-1202 and pembrolizumab (Experimental): All patients will receive TGR-1202 and pembrolizumab. Patients will start receiving TGR-1202 daily for 6 weeks (2 cycles). Pembrolizumab will be given every 3 weeks for 8 cycles. If the daily dose of TGR-1202 (dose level 1) is tolerated in the first cohort the dose will be increased which is the only and final dose escalation. If TGR-1202 is not tolerated the dose will be decreased.
  Interventions: Drug: TGR-1202; Drug: Pembrolizumab

INTERVENTIONS:
Drug: TGR-1202 — TGR-1202 will be given at a dose of 600mg (dose level 1) or 800mg (dose level 2). If the dose of 600mg is tolerated in the first cohort, then the dose will be increased to 800mg which is the only and final dose escalation. If the dose of 600mg is not tolerated, then the dose will be decreased to 400mg daily.
  Other Names: umbralisib
Drug: Pembrolizumab — Pembrolizumab will be given at 200 mg every 3 weeks. The dose will not be adjusted throughout the course of the study.
  Other Names: Keytruda

SUMMARY:
This study will be a standard 3+3 design with a lead in of TGR-1202 at dose of 600mg (dose level 1) or 800mg daily (dose level 2) for 6 weeks, i.e. 2 cycles, followed by pembrolizumab at 200mg every 3 weeks for 8 cycles along with TGR-1202 for patients with relapsed/refractory B-cell NHL or CLL. If the dose of 600mg daily of TGR-1202 (dose level 1) is tolerated in the first cohort the dose will be increased to 800mg qd which is the only and final dose escalation. If TGR-1202 is not tolerated at 600mg daily the dose will be decreased to 400mg daily. The lead in of TGR-1202 was chosen to ensure clinical benefit and to minimize the occurrence of early overlapping toxicity with pembrolizumab as most toxicities were observed early on in the treatment with idelalisib, a related PI3K-inhibitor, and rituximab.

DETAILED DESCRIPTION:
Of note, TGR-1202 has not been associated with treatment related pneumonitis, transaminitis, colitis, PCP-infection nor CMV-reactivation which distinguishes TGR-1202 from idelalisib's toxicity profile.

Once the maximum tolerated dose has been safely reached the study will open an expansion cohort to enroll 18 patients with a patient group in which a clinical signal is detected. Another 7 patients (up to a total of 25 patients in the expansion cohort) may be enrolled after an interim analysis. The duration of therapy will be 2 cycles of TGR-1202 followed by 8 cycles with pembrolizumab and TGR-1202. Thereafter patient will continue on TGR-1202 at the MTD until disease progression. Subjects who experience disease progression while on TGR-1202 maintenance may be eligible for re-treatment with pembrolizumab for up to 6 cycles at the discretion of the Local Investigator if the patient experienced at least disease stabilization during the initial treatment with pembrolizumab, the subject meets the safety parameters listed in the inclusion/exclusion criteria, and the trial is still open. Subjects will resume therapy at the same dose and schedule at the time of initial discontinuation. If safety and feasibility of the combination is confirmed in this dose expansion cohort, a randomized phase II trial comparing TGR-1202 with pembrolizumab versus TGR-1202 could be considered in a larger patient population, possibly within the cooperative group setting for patients with relapsed/refractory B-cell NHL and CLL

The primary objective of the dose expansion cohort will be CR rate. Secondary endpoints will include safety and feasibility, PFS, OS and clinical response (SD, PR, PD).

Patients will be monitored for disease response, adverse events and survival for a minimum of 2 years following enrollment. During and after treatment, patients will be evaluated for toxicities, particularly immunologic adverse events including pneumonitis, autoimmune colitis, dermatitisetc. Peripheral blood, lymph node and bone marrow samples will be collected before and during the treatment course for the correlative studies outlined below. Complete blood counts and differential counts with a complete metabolic panel will be obtained at the time intervals. If the patients are confirmed to have disease progression or intolerable toxicities the patients will be offered alternative treatment at the physicians' discretion. All of the patients will be followed for survival. All patients will receive HSV prophylaxis with acyclovir 400mg po bid or per institutional standards.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Be greater than or equal to 18 years of age on day of signing informed consent.
* Have measurable disease based on iwCLL or Lugano criteria.
* Have had at least 1 prior line of standard therapy
* Be willing to provide tissue from a bone marrow biopsy if suspected involvement and/or lymph node at enrollment, as well, as a repeat bone marrow biopsy (if involved at diagnosis) after 3 of therapy and at the time of progression and/ or completion of therapy whichever comes first.
* Have a performance status of 0-1 on the ECOG Performance Scale.
* Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.

Hematological Absolute neutrophil count (ANC) ≥1000 /mcL Platelets ≥50,000 / mcL (if bone marrow involvement ≥30,000 mcL) Hemoglobin ≥8 g/dL

Renal Serum creatinine OR ≤1.5 X upper limit of normal (ULN) OR Measured or calculateda ≥60 mL/min for subject with creatinine levels > 1.5 X institutional Hepatic ULN creatinine clearance (GFR can also be used in place of creatinine or CrCl)

Hepatic Serum total bilirubin ≤1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤2.5 X ULN Albumin >2.0 mg/dL

Coagulation International Normalized ≤1.5 X ULN unless subject is receiving anticoagulant therapy as Ratio (INR) or long as PT or PTT is within therapeutic range of intended use Prothrombin Time (PT) of anticoagulants

Activated Partial ≤1.5 X ULN unless subject is receiving anticoagulant therapy as Thromboplastin Time long as PT or PTT is within therapeutic range of intended use (aPTT) of anticoagulants

aCreatinine clearance should be calculated per institutional standard.

* Female subject of childbearing potential should have a negative urine or serum pregnancy prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  i. Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

ii. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.

- Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.

Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

* Has a history of non-infectious pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.
* Has received prior therapy with a PI3K-inhibitor. (Prior therapy with a PI3K-inhibitor is allowed if it was discontinued for intolerance)
* Is pregnant or breast feeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of treatment.
* Has known active central nervous system (CNS) disease and/or lymphomatous involvement. Subjects with previously treated CNS lymphoma and/or lymphomatous meningitis may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events | Up to 3 years.
  To determine the maximally tolerated dose of TGR-1202 in combination with pembrolizumab by finding the number of patients with adverse events. This information will be used to determine the recommended phase II dose for this combination for patients with relapsed/refractory CLL/SLL and B-cell NHL.

SECONDARY OUTCOMES:
proportion of patients with complete remission (CR) | Up to 3 years
  The proportion of subjects who achieve a confirmed CR by the the international workshop on CLL (iwCLL) and the Lugano Response Criteria for Non-Hodgkin's Lymphoma.
duration of response (DOR) | Up to 3 years
  The interval from the first documentation of confirmed CR or PR (by IRC) to the first documentation of definitive disease progression or death from any cause. Definitive disease progression is CLL progression based on standard criteria excluding lymphocytosis alone.
progression free survival (PFS) rate | From the start of treatment until the date of first documented progression or date of death from any cause, whichever comes first, up to 100 months
  The interval from the first dose of study drug to the first documentation of definitive disease progression or death from any cause.
MRD negativity rate | Up to 3 years
  The proportion of subjects with MRD <10-4, assessed by flow cytometry in bone marrow.
nodal response rate | Up to 3 years
  The proportion of subjects who achieve a 50% decrease from baseline in the sum of the products of the greatest perpendicular diameters (SPD) of index lesions.
overall survival (OS) rate | From the start of treatment until the date of death from any cause, whichever comes first, up to 100 months
  The interval from the start of study treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Thirman, MD, Principal Investigator — University of Chicago
Locations (3):
- United States (3):
  - Yale University, New Haven, Connecticut
  - University of Chicago, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York